CLINICAL TRIAL: NCT04839627
Title: Impact of Serum Progesterone Levels on the Day of Fresh and Frozen Embryo Transfer on the Ongoing Pregnancy Rates
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Other Study IDs: PROGESTE
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Infertility
Keywords: serum progesterone; embryo transfer; pregnancy rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- serum progesterone measurement
  Interventions: Other: serum progesterone measurement

INTERVENTIONS:
Other: serum progesterone measurement — progesterone levels measurement on the day of the embryo transfer on all AMP cycles

SUMMARY:
Serum progesterone levels prepare the endometrium for implantation and play an important role during embryo transfer (ET). In clinical practice, luteal phase support progesterone supplementation is systematically offered to all women undergoing medically assisted procreation (AMP), independently of ET conditions (fresh and frozen).

The investigators propose to perform a prospective cross-sectional single-center cohort study to measure progesterone levels on the day of the ET on all AMP cycles and to compare these levels between active pregnancies and ET unsuccessful cycles. They will determine progesterone threshold levels corresponding to successful attempts in all ET strategies (fresh and frozen) as well as clinical and biological risk factors leading to luteal phase deficiency during ET. They could therefore individualize progesterone supplementation according to patient's needs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* planned embryo transfer
* signed informed consent

Exclusion Criteria:

* patients falsely included, major inclusion criteria not respected
* lack of social insurance
* refusal to participate in the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who need an embryo transfer in the center.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Serum progesterone levels on the day of embryo transfer | During the procedure
  µg/L

SECONDARY OUTCOMES:
pregnancy rate | 1 month after procedure
  Post-embryo transfer βHCG levels (UI/l).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Joseph Marseille, Marseille, France